CLINICAL TRIAL: NCT02695329
Title: Randomized Controlled Study Comparing Vanguard With KneeAlign2 Navigational System Versus Vanguard Conventional
Brief Title: Vanguard TKA With KneeAlign 2 and Without KneeAlign 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ORTHO.CR.GK53
Record Dates: First submitted 2016-02-19; First posted 2016-03-01 (Estimated); Results first posted 2019-10-03 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-01

CONDITIONS: Osteoarthritis, Knee
Keywords: navigation system; palm-sized; total knee arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vanguard with KneeAlign 2 (Active Comparator): Having total knee arthroplasty surgery with the use of a navigation system KneeAlign 2.
  Interventions: Device: KneeAlign 2
- Vanguard without KneeAlign 2 (No Intervention): Having total knee arthroplasty surgery with the use of conventional surgical instruments, and without a navigation system KneeAlign 2.

INTERVENTIONS:
Device: KneeAlign 2 — Patients suffering non-severe varus deformity Osteoarthritis will be enrolled and randomly assigned into one of two treatment groups. Patients in investigational group will be treated with total knee arthroplasty and the accelerometer-based navigational device. Patients in control group will be treated with total knee arthroplasty with conventional instrumentation.
  Other Names: KneeAlign2
  Arms: Vanguard with KneeAlign 2

SUMMARY:
Purpose of this study is to determine the effectiveness of the KneeAlign 2 system in terms of precise implant alignment by demonstrating that KneeAlign 2 provides better tibial alignment compared to conventional instruments

DETAILED DESCRIPTION:
Purpose of this study is to determine the effectiveness of the KneeAlign 2 system in terms of precise implant alignment by demonstrating that KneeAlign 2 provides better tibial alignment compared to conventional instruments.

ELIGIBILITY:
Inclusion Criteria:

* Knee (either unilateral or bilateral) Osteoarthritis (varus deformity only)
* Subjects willing to return for follow-up evaluations

Exclusion Criteria:

* Knee degenerative diseases other than Knee Osteoarthritis (such as necrosis / Rheumatoid Arthritis)
* Severe OA deformation (FTA: >185 degrees or <175 degrees)
* Active Infection (or within 6 weeks after infection)
* Sepsis
* Osteomyelitis
* Any type of implant is inserted in the affected side of lower extremity
* Hip disease on the affected side
* Uncooperative patient or patient with neurologic disorders who are incapable of following directions
* diagnosed Osteoporosis or Osteomalacia
* Metabolic disorders which may impair bone formation
* Distant foci of infections which may spread to the implant site
* Rapid joint destruction, marked bone loss or bone resorption apparent on roentgenogram
* Vascular insufficiency, muscular atrophy or neuromuscular disease.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-05-24 (Actual); Primary Completion 2018-10-03 (Actual); Study Completion 2018-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yukihide Minoda, Principal Investigator — Osaka City University
Locations (1):
- Osaka City University, Osaka, Japan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vanguard With KneeAlign 2 | Vanguard Without KneeAlign 2
Started | 50 | 50
Completed | 45 | 45
Not Completed | 5 | 5
Not completed — Adverse Event | 1 | 0
Not completed — Poor X-ray quality for measurement | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vanguard With KneeAlign 2 | Vanguard Without KneeAlign 2 | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 4 | 5
  >=65 years | 49 | 46 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.8 (5.2) | 74.0 (6.6) | 74.9 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 40 | 79
  Male | 11 | 10 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 50 | 50 | 100
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 50 | 50 | 100
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.3 (4.2) | 27.3 (4.3) | 26.8 (4.3)
EQ-5D-3L [Mean (Standard Deviation); unit: point] — Measure Description: EQ-5D is patient reported outcome measure to score patient's health related quality of life with minimum score of -0.111 and maximum score of 1.000.
  Higher score means better outcomes. Population: Missing data on 6 KneeAlign group patients and 5 Conventional group patients. Failed to answer all questions on the form.
  point
    number analyzed (Participants) | 44 | 45 | 89
    (all) | 0.553 (0.117) | 0.582 (0.091) | 0.568 (0.105)
KSS-Objective Score [Mean (Standard Deviation); unit: point] — KSS-Objective score is physician-derived component and allows for more than 100 points in patients with greater than 125° of flexion and a stable painless knee as outlined below. Lowest possible score is 0.
  "Alignment" has a maximum of 25 points. "Instability" allows a maximum of 25 points.
  "Joint Motion" allows one point for each 5° of joint motion and allows greater than 25 points for patients with greater than 125° of motion. There are deductions for flexion contracture and extension lag. "Symptoms" category has maximum allowable points 25.
  Higher score means better outcomes. Population: Missing data on 9 KneeAlign2 patients and on 9 Conventional patients. Failed to obtain data.
  point
    number analyzed (Participants) | 41 | 41 | 82
    (all) | 37.4 (19.1) | 35.9 (19.3) | 36.6 (19.1)
KSS-Patient Satisfaction [Mean (Standard Deviation); unit: point] — KSS-Patient Satisfaction is patient-derived score and is a five-question 40-point scale that is collected preoperatively and at each follow-up visit. Lowest possible score is 0.
  Higher score means better outcomes. Population: Missing data, 5 KneeAlign2 patients and 5 conventional patients. Failed to answer all questions on the form.
  point
    number analyzed (Participants) | 45 | 45 | 90
    (all) | 11.2 (6.1) | 13.1 (6.0) | 12.1 (6.1)
KSS-Function Score [Mean (Standard Deviation); unit: point] — KSS-function score is patient-derived score and composed of four subgroups and has a maximum score of 100.
  "Walking and Standing" has a maximum value of 30 points, "Standard Activities" has a maximum of 30 points, "Advanced Activities" has a maximum of 25 points and "Discretionary Activities" has a maximum of 15 points.
  Lowest possible score is 0. Higher score means better outcomes. Population: Missing data on 8 KneeAlign2 patients and 12 Conventional patients. Failed to answer all questions on the form.
  point
    number analyzed (Participants) | 42 | 38 | 80
    (all) | 33.5 (16.5) | 43.6 (18.4) | 38.3 (18.0)
KSS-Patient Expectation [Mean (Standard Deviation); unit: point] — KSS-Patient Expectations is patient-derived score and is a three-question fifteen-point scale that is collected pre-operatively and post-operatively. The pre-operative questions reflect the patient's opinion on the extent to which the patient expects that operation will improve knee pain, and ability to perform activities of daily living and recreational activities. The post-operative questions reflect the extent to which postoperative outcome has met the patient's pre-operative expectations with respect to pain and function.
  The score ranges from 3 to 15. Higher score means better outcomes. Population: Missing data on 16 KneeAlign2 patients and 13 conventional patients. Failed to answer all questions on the form
  point
    number analyzed (Participants) | 34 | 37 | 71
    (all) | 9.1 (2.1) | 9.6 (2.6) | 9.3 (2.4)
Oxford Knee Score [Mean (Standard Deviation); unit: point] — Patient Reported Outcome specific for knee disease. Score range from 0 to 48. Higher score means better outcome. Population: Missing data on 7 KneeAlign2 patients and 3 Conventional patients. Failed to answer all questions on the form.
  point
    number analyzed (Participants) | 43 | 47 | 90
    (all) | 20.7 (8.0) | 24.0 (7.9) | 22.4 (8.1)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects That Have Alignment Within 2 Degrees From Neutral on Tibia
Description: Proportion of subjects that have tibial alignment within 2 degrees from neutral and compare the accuracy of tibial component alignment between two groups.
Time Frame: Postoperative 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Vanguard With KneeAlign 2 | Vanguard Without KneeAlign 2
Number analyzed (Participants) | 45 | 45
Participants
  within 2 degrees (success) | 41 | 31
  outlier (failure) | 4 | 14

2. Secondary Outcome: Number of Participants With Tibial Posterior Slope Alignment Within Predetermined Threshold
Description: Deviation of tibial posterior slope angle from preoperative planned angle (within 2 degrees)
Time Frame: Postoperative 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Vanguard With KneeAlign 2 | Vanguard Without KneeAlign 2
Number analyzed (Participants) | 45 | 45
Participants
  within 2 degrees (success) | 26 | 27
  outlier (failure) | 19 | 18

3. Secondary Outcome: Number of Participants With Femoral Varus/Valgus Angle Within Predetermined Threshold
Description: Deviation of femoral valus/valgus angle from preoperative planned angle (within 2 degrees)
Time Frame: Postoperative 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Vanguard With KneeAlign 2 | Vanguard Without KneeAlign 2
Number analyzed (Participants) | 45 | 45
Participants
  within 2 degrees (success) | 35 | 28
  outlier (failure) | 10 | 17

4. Secondary Outcome: Number of Participants With Adverse Events and/or Adverse Device Effects
Description: Number of participants, who experience adverse events and/or adverse device effects
Time Frame: Intra-operative and Post-operative 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Vanguard With KneeAlign 2 | Vanguard Without KneeAlign 2
Number analyzed (Participants) | 50 | 50
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: From surgery to 6 month visit.
Arm/Group | Vanguard With KneeAlign 2 | Vanguard Without KneeAlign 2
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 1/50 | 0/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vanguard With KneeAlign 2 (N=50) | Vanguard Without KneeAlign 2 (N=50)
Infection (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Postoperative infection

LIMITATIONS AND CAVEATS:
Image assessment, which is primary endpoint, was done on 2D x-ray (not based on CT).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-20): https://cdn.clinicaltrials.gov/large-docs/29/NCT02695329/Prot_SAP_001.pdf